CLINICAL TRIAL: NCT00420732
Title: A Phase II Study of Tergenpumatucel-L (HyperAcute Lung) Cancer Vaccine in Subjects With Advanced Non-Small Cell Lung Cancer Who Responded to First Line Platinum-Doublet Treatment
Brief Title: Vaccine Maintenance Treatment for Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment goals unable to be reached.
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Sponsor
Organization: Lumos Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NLG0201; OBA#0611-820 (Other: Office of Biotechnology Activities)
Record Dates: First submitted 2007-01-08; First posted 2007-01-11 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaccine Group (Experimental)
  Interventions: Biological: HyperAcute-Lung Cancer Vaccine

INTERVENTIONS:
Biological: HyperAcute-Lung Cancer Vaccine — 300 million cells given intradermally every 3 weeks for up to a total of 12 vaccinations
  Other Names: HAL-1, HAL-2, HAL-3

SUMMARY:
To determine the response rate of the administration of HyperAcute-Lung Cancer Vaccine for subjects with stage IIIB or stage IV non-small cell lung cancer who have been treated with first line platinum-doublet therapy and have responded or are considered to have stable disease.

DETAILED DESCRIPTION:
Unfortunately, despite the best clinical efforts and breakthroughs in biotechnology, most patients diagnosed with advanced stage lung cancer continue to die from their disease. Reasons for this include that: 1) patients are often diagnosed at a time when their lung cancer has already spread to other sites such as the chest cavity, bone, lung, liver, and brain limiting the options for local radiation therapy and surgery, and 2) the cancer cells are resistant or become resistant to chemotherapy drugs used to treat the patient. Resistance to one type of chemotherapy agent often rapidly leads to resistance against many other chemotherapy drugs.

These reasons are the major causes of cancer progression that are usually discussed when considering treatment options for patients with disease that continues to grow and spread. However, another important part of the body should be considered-- the immune system. Scientists have clearly shown that lung cancer cells produce a number of abnormal proteins or abnormal amounts of certain proteins found in normal lung cells. Normally one would expect a patient to develop an immune response against these abnormal proteins found in their cancer and attack them much the way we would fight off an infection from a foreign bacteria or virus. However, for reasons that scientists do not fully understand, the immune system fails to respond to these abnormal proteins and does not attack the lung cancer cells. This human clinical trial proposes a new way to make the immune system recognize the cancer and encourage it to attack the cancer cells.

Many people are familiar with the idea of transplants between people of organs like the kidneys or heart. When an organ transplant between two people is completed one of the problems that can occur is rejection of the donated organ by the recipient. This can occur because the immune system of the patient who receives the organ attacks the donated organ. If you were to attempt to transplant a pig heart to a human the rejection would be dramatically stronger than when organs are transplanted between two people. This is partly because lower animals express sugar-protein patterns on the surface of their cells that humans do not. In fact, our immune systems can quickly recognize tissues from lower mammals such as the pig or the mouse and destroys them.

In this project, we have put a mouse gene into human lung cancer cells that produces these abnormal sugar patterns and stimulates the immune system to attack the lung cancer. This strategy works well to kill human other cancer cells in the laboratory, but it needs to be tried in lung cancer patients to see if it will be effective and to determine if such a treatment causes any side effects. We propose to test this new treatment in subjects with non-small cell lung cancer to see if it can stop, slow or destroy tumors in these subjects. Subjects will be injected with an anti-tumor vaccine consisting of a mixture of three types of dead human lung cancer cells that have been genetically altered to express the mouse gene responsible for making this abnormal sugar-protein on the cells.

ELIGIBILITY:
Inclusion Criteria:

* histological diagnosis of non-small cell lung cancer. Squamous cell (epidermoid), adenocarcinoma, bronchoalveolar carcinoma and large cell anaplastic lung carcinoma histologies are eligible. Mixed NSCLC/small cell, and variant large and small are not eligible.
* AJCC Stage IIIB(pleural effusion) or Stage IV NSCLC
* Subjects must have been previously treated with only a first line platinum-doublet therapy that may or may not include Avastin(R). Those treated with definitive chemo-radiation with curative or palliative intent or who have received multiple regimens are not eligible.
* Subjects' NSCLC must have responded or remained stable through first line platinum-doublet therapy.
* ECOG Performance Status ≤ 2.
* Serum albumin ≥ 3.0 gm/dL.
* Expected survival ≥ 6 months.
* Hemoglobin ≥ 9.0 g/dl
* Platelets ≥ 100,000 cells/mm3
* ANC ≥ 1500 cells/mm3
* Serum total bilirubin ≤ 2 x ULN, ALT and AST ≤ 2.5 x ULN (≤5 if hepatic metastasis is present).
* Serum creatinine ≤ 1.5 x ULN, or creatinine clearance ≥ 50 ml/min.
* Measurable or non-measurable disease.
* Subjects must have negative serology for HIV prior to entering study.
* Male and female subjects of child bearing potential must agree to use contraception or avoidance of pregnancy measures while enrolled on study and receiving experimental drug, and for one month after the last immunization.

Exclusion Criteria:

* Age < 18 years.
* Active CNS metastases or carcinomatous meningitis.
* Subjects' whose NSCLC progressed during/after first line platinum-doublet therapy.
* Subjects having undergone splenectomy.
* Hypercalcemia > 2.9 mmol/L, unresponsive to standard therapy.
* Pregnant or nursing women.
* Other malignancy within the last 5 years, unless the probability of recurrence of the prior malignancy is < 30%. Patient's curatively treated for squamous and basal cell carcinoma of the skin and carcinoma in situ of the uterine cervix (CIN) or subjects with a history of malignant tumor in the past that have been disease free for at least five years are also eligible for this study.
* History of organ transplant.
* Current, active treatment with immunosuppressive therapy such as cyclosporine, tacrolimus, etc.
* Subjects taking systemic corticosteroid therapy for any reason including replacement therapy for hypoadrenalism, are not eligible. Subjects receiving inhaled or topical corticosteroids are eligible.
* Significant or uncontrolled congestive heart failure, myocardial infarction, significant ventricular arrhythmias within the last six months or significant pulmonary dysfunction.
* Active infection or antibiotics within 1-week prior to study, including unexplained fever.
* Autoimmune disease.
* Any condition, psychiatric or otherwise, that would preclude informed consent, consistent follow-up or compliance with any aspect of the study.
* A known allergy to any component of the vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-01; Primary Completion 2012-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To determine the response rate of the administration of HyperAcute® Lung (HAL) Cancer Vaccine cells by injection into subjects with stage IIIB (pleural effusion) or stage IV non-small cell lung carcinoma who have been treated with first line platinum-dou | 4 months

SECONDARY OUTCOMES:
To conduct correlative scientific studies of subject samples to determine the mechanism of any observed antitumor effect. In these studies human humoral and cellular immune responses to HAL cells will be evaluated. | while on study

CONTACTS AND LOCATIONS:
Overall Officials: Charles J. Link, Jr., M.D., Study Chair — NewLink Genetics Corporation
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Washington University in St. Louis, St Louis, Missouri